CLINICAL TRIAL: NCT05863312
Title: Rhegmatogenous rEtinal Detachment With or withOut Scleral Buckle (REDOS) Trial: a Factorial, Randomized Controlled Trial
Brief Title: REtinal Detachment Outcomes Study
Acronym: REDOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Fighting Blindness Canada (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-6508
Record Dates: First submitted 2023-05-08; First posted 2023-05-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Retinal Detachment
Keywords: Pars plana vitrectomy; Scleral buckle; Rhegmatogenous retinal detachment; Proliferative vitreoretinopathy; Anatomic success; Visual acuity; Retinal displacement; Postoperative pain; Quality of life; Complications
MeSH Terms: conditions — Retinal Detachment; Vitreoretinopathy, Proliferative; Pain, Postoperative | interventions — Scleral Buckling; perflutren

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pars plana vitrectomy + sulfur hexafluoride gas tamponade (Active Comparator)
  Interventions: Procedure: Pars plana vitrectomy; Other: Sulfur hexafluoride gas tamponade
- Pars plana vitrectomy with scleral buckle + sulfur hexafluoride gas tamponade (Experimental)
  Interventions: Procedure: Pars plana vitrectomy with scleral buckle; Other: Sulfur hexafluoride gas tamponade
- Pars plana vitrectomy + perfluoropropane gas tamponade (Experimental)
  Interventions: Procedure: Pars plana vitrectomy; Other: Perfluoropropane gas
- Pars plana vitrectomy with scleral buckle + perfluoropropane gas tamponade (Experimental)
  Interventions: Procedure: Pars plana vitrectomy with scleral buckle; Other: Perfluoropropane gas

INTERVENTIONS:
Procedure: Pars plana vitrectomy — Pars plana vitrectomy will be performed in a standard fashion starting with central vitrectomy, then by localizing retinal breaks, and marking them with endodiathermy. Perfluorocarbon will be used to displace subretinal fluid which will be aspirated at its exit from the retinal break as much as possible and maximal vitreous base shaving will be performed in all cases. This will be followed by an air-fluid exchange. Use of cryotherapy to solidify the retina intraoperatively and use of internal limiting membrane peeling of the posterior pole will be at the discretion of the surgeon. In all cases, laser photocoagulation around retinal breaks, holes, areas of lattice degeneration, and posterior to sclerotomy sites will be done and then a 360° laser retinopexy will be performed at the surgeon's discretion and consisted of three rows of medium-white burns anterior to the level of the vortex vein, towards and beyond the equator.
  Other Names: PPV
  Arms: Pars plana vitrectomy + perfluoropropane gas tamponade; Pars plana vitrectomy + sulfur hexafluoride gas tamponade
Procedure: Pars plana vitrectomy with scleral buckle — In cases with SB, after 360° peritomy and dissection in 4 quadrants, a 41-circling band with 3082 sleeves (Labtician Ophthalmics, Oakville, ON Canada) will be used in all cases and fixed to the sclera at approximatively 11.5 mm from the limbus (or 5.5 from the insertion of rectus muscles) using partial thickness scleral tunnel or mattress sutures with 5.0 prolene or nylon performed in 4 quadrants depending on the surgeon preferences. Pars plana vitrectomy will then be performed as in the PPV only group.
  Other Names: PPV-SB
  Arms: Pars plana vitrectomy with scleral buckle + perfluoropropane gas tamponade; Pars plana vitrectomy with scleral buckle + sulfur hexafluoride gas tamponade
Other: Sulfur hexafluoride gas tamponade — At the end of the surgery, the eye is filled with sulfur hexafluoride gas tamponade.
  Other Names: SF6
  Arms: Pars plana vitrectomy + sulfur hexafluoride gas tamponade; Pars plana vitrectomy with scleral buckle + sulfur hexafluoride gas tamponade
Other: Perfluoropropane gas — At the end of the surgery, the eye is filled with perfluoropropane gas tamponade.
  Other Names: C3F8
  Arms: Pars plana vitrectomy + perfluoropropane gas tamponade; Pars plana vitrectomy with scleral buckle + perfluoropropane gas tamponade

SUMMARY:
Background: Few large randomized controlled trials provide strong evidence to guide surgical repair of primary rhegmatogenous retinal detachment (RRD) repair. The purpose of this factorial, single-blind, randomized controlled trial is to analyze and compare the surgical outcomes, functional visual outcomes, complications, and quality of life associated with RRD repair using (A) pars plana vitrectomy only (PPV) or PPV with scleral buckle (PPV-SB) and (B) sulfur hexafluoride gas (SF6) or perfluoropropane gas (C3F8) tamponade.

Methods: Eligible patients with moderately complex RRD will be randomized 1:1 to PPV or PPV-SB and 1:1 to SF6 or C3F8 gas tamponade. Approximately 560 patients will be recruited to be able to detect a difference of around 10% in SSAS rate between groups. Patients will be followed using multimodal imaging and quality of life questionnaires before and after the surgical repair until 1 year postoperative. The primary outcome will be single surgery anatomic success (SSAS), defined as absence of reoperation for recurrent RRD in the operating room. Secondary outcomes will be pinhole visual acuity (PHVA) at 8-10 weeks and 6 months, final best-corrected visual acuity (BCVA), final retina status (i.e., attached or detached), time to onset of RRD recurrence, severity and number of complications, and questionnaire results.

Discussion: This will be the first 2 × 2 factorial randomized controlled trial examining repair techniques in primary RRD. It will also be the first randomized controlled trial to compare gas tamponade between the two most common agents. Notably, it will be adequately powered to detect a clinically significant effect size. The use of multimodal imaging will also be a novel aspect of this study, allowing us to compare head-to-head the impact of adding an SB to the retina's recovery after RRD repair and of differing gas tamponades. Until now, the treatment of RRD has been largely guided by pragmatic retrospective cohort studies. There is a lack of strong evidence guiding therapeutic decisions and this trial will address (1) whether supplemental SB is justified and (2) whether longer duration gas tamponade with C3F8 is necessary.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosis of rhegmatogenous retinal detachment

Exclusion Criteria, retinal detachment with:

* Proliferative vitreoretinopathy (PVR) grade ≥C2
* Chronic RRD with duration >3 months
* Proliferative diabetic retinopathy with tractional retinal detachment (RD)
* Macular holes
* Epiretinal membrane grade 3 or 4
* Traumatic RD
* Giant retinal tears
* Retinal dialysis
* Foveoschisis
* Wet age-related macular degeneration
* Endophthalmitis
* Acute retinal necrosis
* Coats disease
* Retinopathy of prematurity
* Retinoschisis
* Retinal colobomas
* Prior glaucoma surgery or strabismus surgery (favoring PPV only)
* Superior RD extent less than 3 clock hours (favoring PPV only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2023-09-26 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Single surgery anatomic success | Until final 1 year follow-up
  Freedom from reoperation for recurrent RRD

SECONDARY OUTCOMES:
Pinhole visual acuity | 8-10 weeks, 6 months
Best-corrected visual acuity | 1 year
Time to onset of RD recurrence | Until final 1 year follow-up
Severity and number of complications | Until final 1 year follow-up
Quality of life questionnaire | 2 weeks, 8-10 weeks, 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ali Dirani, MD MSc MPH, Principal Investigator — CHU de Québec - Université Laval; Mélanie Hébert, MD MSc, Principal Investigator — CHU de Québec - Université Laval
Locations (1):
- Hôpital du Saint-Sacrement, CHU de Québec - Université Laval, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
The full protocol will be published in the journal Trials. The final trial dataset could be made available to other research teams upon reasonable request and after evaluation of the request by the trial team. The shared dataset will be coded and will not include any identifying patient data.

REFERENCES:
- [Derived] Hebert M, Bourgault S, Caissie M, Tourville E, Dirani A. REtinal Detachment Outcomes Study (REDOS): study protocol for a factorial, randomized controlled trial. Trials. 2023 Dec 20;24(1):820. doi: 10.1186/s13063-023-07815-x. PMID 38124155